CLINICAL TRIAL: NCT01052337
Title: Anesthesia Induction With Propofol or Sevoflurane in Patients Undergoing Fiberoptic Intubation for Cervical Myelopathy: Effects on Heamodynamics
Brief Title: Anesthesia Induction in Patients Undergoing Surgery for Cervical Myelopathy
Acronym: Blade runner
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Federico Bilotta, Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Blade-runner
Record Dates: First submitted 2010-01-12; First posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-12

CONDITIONS: Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator)
  Interventions: Drug: anaesthetics: sevofluorane
- sevofluorane (Active Comparator)
  Interventions: Drug: anaesthetics: sevofluorane

INTERVENTIONS:
Drug: anaesthetics: sevofluorane — 0.5%of sevofluorane with air

SUMMARY:
Aim of this trial is to compare propofol-based anaesthesia vs. sevoflurane-based anaesthesia induction in patients with cervical myelopathy receiving oral or nasal fiberoptic intubation.

DETAILED DESCRIPTION:
Background: Fiberoptic intubation is the preferred method of intubation in patients with acute symptoms or signs of cervical myelopathy. This approach minimizes cervical spine movements to prevent new neurologic deficits or further neurologic injury, and is the safer method to secure the airways in patients with foreseen difficult intubation. In these patients anaesthesia induction is aimed to prevent cervical spine movements and to maintain hemodynamic stability. The most commonly reported technique for anaesthesia induction in patients with cervical myelopathy is based on local anaesthesia and propofol administration. Aim of this trial is to compare propofol-based anaesthesia vs. sevoflurane-based anaesthesia induction in patients with cervical myelopathy receiving oral or nasal fiberoptic intubation.

Methods: This randomized controlled trial is designed to prove equivalence. A series of 116 patients aged between 18 and 75 years, with cervical myelopathy will be enrolled. In all patients topical anaesthesia will be accomplished before anaesthesia induction. Patients will be randomly assigned to one of two anaesthesia induction strategies (sevoflurane + O2 + air or propofol + O2 + air). When loss of consciousness occurs (indicated by Bispectral index values between 40 and 50), oral or nasal fiberoptic intubation will be performed. The hemodynamic effects of the anaesthesia induction strategies will be assessed measuring mean arterial pressure at 4 time points: before anaesthesia induction (T1: baseline), at the end of anaesthesia induction when an adequate sedation level, with Bispectral index values 40-50, is achieved (T2: sedation steady state); immediately after placement of endotracheal tube (T3: intubation); five minute after tracheal intubation (T4: post-intubation). Secondary end-points of the study include the incidence of apnoea during induction process, diagnosed as absence of carbon dioxide trace for more than 10 seconds, the incidence of induction complications, defined as presence of laryngospasm, coughing and patient movement, and intubation conditions, defined as cord opening.

Discussion: We present the development phase of this anaesthesiological trial. A total of 40 patients have been enrolled from April 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing cervical spine surgery;
* Male or female;
* Aged 18-75 years.

Exclusion Criteria:

* Severe cardiovascular pathology;
* Liver disease;
* Renal disease;
* BMI >35;
* Allergies to any anaesthetic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
episode of severe arterial hypotension | at 0 minut, after 3 minuts, after 5 minuts

SECONDARY OUTCOMES:
the incidence and duration of apnoea and the incidence of induction complications such as laryngospasm, coughing and patient movement during fiberoptic intubation. | at 0 minuts , at 5 minuts

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico UMBERTO I, Rome, Rome, Italy